CLINICAL TRIAL: NCT00435903
Title: Pilot Study of the Feasibility of Palm Pilots in Monitoring Smoking Behavior in Individuals With Chronic Mental Illness
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North Suffolk Mental Health Association (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CORRC #21-04
Record Dates: First submitted 2007-02-14; First posted 2007-02-16 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2007-02

CONDITIONS: Smoking
Keywords: smoking; self-monitoring; major mental illness; palm pilots; subjects with DSM-IV Axis I diagnosis
MeSH Terms: conditions — Smoking

INTERVENTIONS:
Device: Palm Pilot

SUMMARY:
The goal of this open trial is to pilot the use of palm pilots as a tool for monitoring smoking behavior in individuals with serious mental illness. That is, the investigators aim to assess the usefulness and feasibility of using Palm Pilots as a tool for monitoring smoking behavior and for coaching participants to use a strategy for delaying and reducing cigarette use.

DETAILED DESCRIPTION:
The specific aims of this project are:

1. We will compare the accuracy of daily palm pilot recordings to paper and pencil measures. We hypothesize that the number of cigarettes smoked according to daily palm pilot recordings will correlate as well with salivary cotinine levels (a metabolite of nicotine) as will daily paper and pencil recordings. That is, we expect that palm recordings will be as accurate as paper and pencil recordings.
2. We will compare the total number of smoked cigarettes reported by the daily ratings (paper and pencil or palm pilot) to participants' report of their weekly totals. We expect that participants will tend to underestimate the number of cigarettes smoked when asked to report weekly totals. That is, we hypothesize that participants will report smoking fewer cigarettes in their weekly total compared to their daily reports of smoking and that totals based on daily reports will correlate more strongly with cotinine levels.
3. We will measure the frequency at which participants access a screen on the Palm Pilot that presents the "4 D's," which are four strategies for delaying or reducing cigarette use. Participants will be asked to access this screen when they experience an urge to smoke. We hypothesize that at least some participants will make use of this screen.
4. We will assess the effect of daily monitoring on salivary cotinine levels. Smoking reduction is not a specific goal of this program. However, participants who access the 4D's coaching screen on the Palm when they have an urge may reduce their smoking. We hypothesize that reduction in cotinine levels will be correlated with greater frequency of accessing the 4 D's screen. That is, participants who access the 4D's screen most often (more than 5 times per day) are expected to show more reduction in cotinine levels compared to baseline than are participants who do not access the 4 D's screen
5. We will measure participants' level of satisfaction with the Palm Pilot and the paper and pencil versions of the monitoring forms. We hypothesize that participants will report high levels of satisfaction with the Palm Pilot version, and that these will be as high as or higher than levels of satisfaction with the paper and pencil version.
6. We will assess whether participants are able to complete a rating scale on the Palm Pilot. We hypothesize that participants will be able to complete this scale.
7. We will assess the amount of training time required to train participants to use either the paper and pencil or Palm Pilot versions of the monitoring form.

Methods and Procedures: Ten participants will come in for four, 45-minute assessments, for a total of 3 hours, over a 3-week period. At each visit, smoking behavior will be assessed using either the palm pilot or paper and pencil recordings and carbon monoxide and salivary cotinine will be measured. Training will be provided in the use of the palms and participants will do a "trial" recording of data before their actual data are recorded. In addition, during each week in which participants use Palm Pilots, they will be asked to come into the clinic for a mid-week visit to have their Palm Pilot charged and synced with the computer. No assessments will be completed during these mid-week visits.

Subjects will serve as their own controls in the study. Participants will be asked to keep track of their smoking and to answer questions about their smoking using two formats: paper and pencil forms and forms programmed on Palm Pilots. For the Palm Pilot recordings, participants will be loaned a Palm Pilot to use to answer questions about their smoking whenever they smoke. Palm recordings and paper and pencil recordings will be compared to salivary cotinine and carbon monoxide levels. To control for the effects of one data collection strategy being used before the other, subjects will be randomized to do either paper and pencil recordings or palm recordings first. We will also teach clients a basic behavioral strategy ("the four D's") for cutting down on the amount of cigarettes smoked. The four D's stand for 1) deep breathing, 2) drink fluids, 3) delay, and 4) do something else. The paper and Palm Pilot versions of the questionnaires will include a reminder about the four D's to encourage participants to cut down on the amount of cigarettes smoked per day. In addition, participants will be asked to fill out the Hughes-Hatsukami Scale, which is a measure of nicotine withdrawal symptoms.

In summary, all participants will take part in the following:

1. Assessment 1: Baseline assessment (week 0) will include self report of cigarettes smoked in the past week, a measure of salivary cotinine level, and expired air carbon monoxide level. The four D's strategy for cutting down number of cigarettes smoked will be introduced.
2. For Week 1, subjects will be asked to keep daily paper-and-pencil records of their smoking behavior for the week following baseline. Subjects will be asked to report on number of cigarettes smoked, time of day smoked, how they felt when they smoked, and the degree to which they craved the cigarette. They will also be asked to indicate whether or not they tried any of the four D's strategies to avoid or delay smoking. Additionally, they will fill out the Hughes-Hatsukami Scale once per day.
3. Assessment 2: Subjects will then return for assessment at the end of the week of paper and pencil recordings. Salivary cotinine and carbon monoxide levels will be measured at this time. Additionally, subjects will fill out a satisfaction questionnaire regarding their satisfaction with the paper-and-pencil method of monitoring their smoking.
4. Subjects will be trained to record their smoking behavior using a Palm Pilot version of the recording form. Subjects will be loaned a Palm Pilot that will be programmed to present a computerized version of the smoking behavior monitor form that was used to make paper and pencil recordings. Subjects will be asked to hit a button on the Palm Pilot whenever they have an urge to smoke, and to complete the recordings on the Palm Pilot in the same manner as they did with paper-and-pencil recordings. However, Palm Pilots will be set to beep 1x per day (participant's stated wake-up time) to prompt participants to make a summary recording of number of cigarettes per day and to complete the Hughes-Hatsukami Scale. Additionally, the morning questionnaire will include a reminder screen that encourages participants to make the recordings and to practice the four D's. Subjects will practice using the Palm Pilot over Week 2.
5. Mid-week visit 1: Participants will return to the clinic during the middle of the week to charge and hot-sync (synchronize with the computer) their Palm Pilot. No assessments will occur during this visit.
6. Assessment 3: Subjects will return after a week of practice. Salivary cotinine and carbon monoxide levels will be measured, as well as smoking withdrawal symptoms.
7. Subjects will then be asked to record their smoking on the palm pilots for another week (Week 3).
8. Mid-week visit 2: Participants will return to the clinic during the middle of the week to charge and hot-sync (synchronize with the computer) their Palm Pilot. No assessments will occur during this visit.
9. Assessment 4: Subjects will return for a fourth and final assessment of cotinine and carbon monoxide levels. Subjects will also complete a satisfaction questionnaire regarding their experience with using the Palm Pilot version of monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50
2. Having a DSM-IV psychiatric diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, or major depression with significant functional impairment
3. Smoking 10 or more cigarettes per day
4. Having an expired air minimum CO of at least 10 ppm
5. Normal or corrected to normal eyesight and adequate manual dexterity to operate a palm pilot (will be assessed on case by case basis with participants completing an initial screening which involves demonstrating basic ability to read the screen on the palm pilot and operate the stylus)
6. Stable psychiatric symptoms

Exclusion Criteria:

1. Mini Mental State exam score less than 24/30
2. Currently using nicotine replacement therapy
3. Diagnosis of dementia, neurodegenerative disease, substance abuse or dependence disorders (to substances other than nicotine) active within the last 3 months
4. Patients who, in the investigator's opinion, pose a current homicide or suicide risk

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11
Dates: Start 2005-06; Study Completion 2005-10

PRIMARY OUTCOMES:
We will compare palm-recordings with paper and pencil recordings to examine how well these correlate.

SECONDARY OUTCOMES:
Correlations will be used to compare the total number of smoked cigarettes reported by the daily ratings (paper and pencil or palm pilot) to participants' report of their weekly totals.
We will measure the frequency at which participants access a screen on the Palm Pilot that presents the "4 D's," which are four strategies for delaying or reducing cigarette use.
Repeated measured t-tests will be used to compare participants' cotinine levels before and after participating in this program.
We will use an independent samples t-test to compare satisfaction scores for the two monitoring methods.
We will assess the degree of compliance with completing the mood rating scale (how many out of 7 were completed in the week) and will compare compliance rates for the Palm and paper-and-pencil versions using an independent samples t-test.
We will assess the amount of training time required to train participants to use either the paper and pencil or Palm Pilot versions of the monitoring form.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Friedman-Yakoobian, Ph.D., Principal Investigator — Freedom Trail Clinic
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States